CLINICAL TRIAL: NCT02137720
Title: Translating Telephonic Diabetes Self-management Support to Primary Care Practice: The NYC Care Calls Trial
Brief Title: Translating Telephonic Diabetes Self-management Support to Primary Care Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Jeffrey Gonzalez, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-422; 1R18DK098742-01A1 (NIH)
Record Dates: First submitted 2014-05-08; First posted 2014-05-14 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Treatment Adherence; Self-management; Emotional Distress; Diabetes-related Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephonic Diabetes Self-Management Support (Experimental): This group receives all the Educational Print Materials received by the comparison condition plus telephone calls from a health educator to provide tailored diabetes self-management training and support. Participants with significant emotional distress at baseline also receive additional calls focused on distress management.
  Interventions: Behavioral: Telephonic Diabetes Self-Management Support
- Educational Print Materials (Active Comparator): Participants randomized to this arm will receive print materials on diabetes, glycemic control, self-management, and distress/depression.
  Interventions: Other: Educational Print Materials

INTERVENTIONS:
Behavioral: Telephonic Diabetes Self-Management Support
  Arms: Telephonic Diabetes Self-Management Support
Other: Educational Print Materials
  Arms: Educational Print Materials

SUMMARY:
The goal of this study is to evaluate the implementation and effectiveness of an intervention to improve diabetes self-management, emotional distress and metabolic control among adults with type 2 diabetes receiving care in primary care practices throughout New York City. The program will be implemented by the New York City Department of Health, through their Primary Care Improvement Project.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Receiving treatment for diabetes at selected primary care practices throughout New York City
* Most recent HbA1c ≥ 7.5% (max 3 months prior to randomization)
* Ability to speak and read English or Spanish (or someone in the household who will read to them)
* Access to a telephone
* Willing to give informed consent to participate and accept random assignment.

Exclusion Criteria:

* Stated intention to move out of the New York City area during the next year
* Mental incapacity (e.g., confusion) evident on first telephone contact by Department of Health staff
* Treatment provider deems that the patient is inappropriate for the trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline at 12 months
  Obtained from electronic medical record.

SECONDARY OUTCOMES:
Diabetes Self-Management | Change from baseline at 12 months
  Measured by self-report questionnaire
Medication Adherence | Change from baseline at 12 months
  Measured by self-report questionnaire
Diabetes-related distress | Change from baseline at 12 months
  Measured by self-report questionnaire
Depressive symptoms | Change from baseline at 12 months
  Measured by self-report questionnaire
Blood pressure | Baseline and 12 months
  Obtained from electronic medical record.
Cholesterol | Baseline and 12 months
  Obtained from electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gonzalez, PhD, Principal Investigator — Albert Einstein College of Medicine; Winfred Y Wu, MD, MPH, Principal Investigator — New York City Department of Health and Mental Hygiene
Locations (1):
- New York City Department of Health and Mental Hygiene, New York, New York, United States

REFERENCES:
- [Derived] Gonzalez JS, Hoogendoorn CJ, Linnell J, Fishman S, Jonas V, Pham-Singer H, Schechter CB, Walker EA, Wu WY. Design and methods of NYC care calls: An effectiveness trial of telephone-delivered type 2 diabetes self-management support. Contemp Clin Trials. 2020 Nov;98:106166. doi: 10.1016/j.cct.2020.106166. Epub 2020 Oct 3. PMID 33022367